CLINICAL TRIAL: NCT06979037
Title: Clinical Investigation of Genetic Markers in Diabetic Ulcers and Their Role in Personalized Treatment Targeting
Brief Title: Genetic Markers of Diabetic Ulcers and Personalized Treatment Targets Research
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of University of South China (Other)
Responsible Party: Sponsor
Other Study IDs: NHFY20240506
Record Dates: First submitted 2025-05-05; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Diabetic Ulcers
Keywords: Diabetic Ulcers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood, ulcer tissue, and fecal samples from diabetic ulcer patients will be collected and detected.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This clinical trial involves collecting peripheral blood, ulcer tissue, and fecal samples from diabetic ulcer patients for bioinformatics analysis to screen genetic markers significantly associated with ulcer risk and healing differences. Furthermore, multi-omics data will be integrated to establish a diabetic ulcer risk prediction model. Based on key single nucleotide polymorphisms and their regulatory pathways, potential new drug targets for promoting healing will be explored, providing a genetic basis for personalized treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1) Subjects who voluntarily participate in this clinical study and sign informed consent;
* 2) Patients with type 2 diabetes and diabetic ulcers;
* 3) Disease duration ≥ 10 years or age ≥ 55 years at enrollment;
* 4) Inpatient or outpatient who can be monitored by the same investigating team throughout the duration of the study.

Exclusion Criteria:

* 1) Severe vascular occlusion or impairment;
* 2) Patients with congenital heart disease, aortic dissection, or other severe cardiovascular diseases;
* 3) Patients with ulcers caused by factors other than diabetes;
* 4) Patients with severe liver and kidney dysfunction or serious neurological impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of diabetic ulcer patients who visit the The First Affiliated Hospital of University of South China during the trial period and meet the inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 712 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2027-05-16 (Estimated); Study Completion 2027-05-16 (Estimated)

PRIMARY OUTCOMES:
Ulcer Healing Time | Three years

SECONDARY OUTCOMES:
Absolute Change in Ulcer Area | Three years
  Absolute change in ulcer area over three years in cm2
Number of Amputation Events | Three years
Ulcer Recurrence | Three years
  Number of diabetic foot ulcers with recurrence at three years
Time to Complete Wound Closure | Three years or wound closure
  Time to 100% wound closure utilizing Cox proportional hazards model, a statistical measure of difference of time to event (healing). The analysis will consider covariates that might influence the outcome in the trial.
Number of Foot Infections | Three years
Quality of Life Assessment | Three years
  The Cardiff Wound Impact Schedule questionnaire to measure quality of life. Measure of well-being items from each scale are summated, physical symptoms, everyday living and social life. The items are rated for the extent of the experience and each item is given a number value. This allows the patients to weight the items included in the scale. The well-being scale is scored on a 5-point Likert scale, with response options from 'strongly agree' to 'strongly disagree'. All three scales are then transformed onto a minimum = 0 up to a maximum = 100, where a low score indicates worse, and a high score indicates better feeling of well-being.
Length of Stay | Three years

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of University of South China, Hengyang, Hunan, China

IPD SHARING:
Plan to Share IPD: No